CLINICAL TRIAL: NCT05546723
Title: LUMT1A22, Phase 1 Study of BAFF CAR T Cells (LMY-920) for Treatment of Relapsed or Refractory Myeloma (LMY-920-002)
Brief Title: LMY-920 for Treatment of Relapsed or Refractory Myeloma
Acronym: LMY-920-002
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Luminary Therapeutics (Industry)
Collaborators: The Cleveland Clinic (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LMY-920-002; LUMT1A22 (Other: Cleveland Clinic Taussig Cancer Institute)
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma, Refractory; Multiple Myeloma in Relapse
Keywords: multiple myeloma; CAR-T; BAFF ligand
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Open label, dose escalation study with up to four dose levels of LMY-920. The maximum tolerated dose (MTD) of LMY-920 will be determined using dose-escalation 3+3 design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LMY-920 dose escalation (Experimental): Open label, dose escalation study with up to four dose levels of LMY-920. The maximum tolerated dose (MTD) of LMY-920 will be determined using dose-escalation 3+3 design.
  Interventions: Biological: Autologous CAR-T cell therapy expressing the BAFF-ligand.

INTERVENTIONS:
Biological: Autologous CAR-T cell therapy expressing the BAFF-ligand. — LMY-920

SUMMARY:
Since CAR-T cell treatment of refractory myeloma has shown success, based on preclinical data, we posit that CAR-T cells expressing B-cell activating factor (BAFF) can become another strategy to treat refractory myeloma, even after relapse following BCMA targeting CAR-T cell treatment. This will be phase 1 study of BAFF ligand CAR-T cells in relapsed and refractory myeloma.

DETAILED DESCRIPTION:
In this open label, dose escalation study, up to four dose levels of autologous BAFF ligand CAR-T cells (LMY-920) will be evaluated for treatment relapsed and refractory myeloma. BAFF receptor family includes B-cell activating factor receptor (BR3), B-cell maturation antigen (BCMA) and transmembrane activator and calcium modulator and cyclophilin ligand interactor (TACI). The maximum tolerated dose (MTD) of LMY-920 will be determined using dose-escalation 3+3 design. The primary goal of this study is to determine recommended phase II dose of human LMY-920 in patients with relapsed or refractory myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically confirmed myeloma relapsed or refractory after 3 or more lines of therapy including an immunomodulatory agent, a proteasome inhibitor and an anti-CD38 antibody. Failing line of therapy is defined accordingly to International Myeloma Workshop Consensus Panel.
2. No evidence of CNS myeloma.
3. Male or female > 18 years of age.
4. ECOG Performance status ≤ 2.
5. Has measurable disease at the time of enrollment as defined by at least one of the following:

   * Serum M-protein greater or equal to 0.5g/dL
   * Urine M-protein greater or equal to 200mg/24hr
   * Serum free light chain (FLC) assay: involved light chain greater or equal to 10mg/dL provided serum FLC ratio is abnormal
   * Bone marrow plasma cells greater than or equal to 30% total bone marrow cells
6. >2 weeks since prior radiation therapy or systemic therapy at the time of leukapheresis.
7. Total bilirubin ≤ 1.5 mg/dL (except in patients with Gilbert's syndrome).
8. AST (SGOT)/ALT ≤ 2.5 X institutional upper limit of normal.
9. Serum creatinine < 2 mg/dL.
10. Cardiac ejection fraction of >45%, and no evidence of pericardial effusion, as determined by an echocardiogram.
11. Adequate pulmonary function as defined as pulse oximetry ≥ 92% on room air.
12. Subjects (or legal guardians) must have the ability to understand and the willingness to sign a written informed consent document.
13. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 90 days after the BAFF CAR-T cell infusion.
14. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

1. ASCT within 6 weeks of informed consent.
2. History of allogeneic hematopoietic stem cell transplantation.
3. Active graft-versus-host disease.
4. Active central nervous system or meningeal involvement by myeloma. Subjects with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of CNS or meningeal involvement must be in a documented remission by CSF evaluation and contrast-enhanced MRI imaging for at least 90 days prior to registration.
5. Active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast).
6. Less than 28 days elapsed between prior treatment with investigational agent(s) and the day of lymphocyte collection.
7. New York Heart Association class IV congestive heart failure.
8. Cardiovascular disorders including unstable angina pectoris, clinically significant cardiac arrhythmias, myocardial infarction or stroke (including transient ischemic attack, or other ischemic event) within 6 months prior to registration.
9. Active infection requiring intravenous systemic treatment.
10. HIV seropositivity.
11. Pregnant or breastfeeding women are excluded from this study because LMY-920 therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with LMY-920, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
12. Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy.
13. Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.)
14. Patients with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.
15. Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
16. Known additional malignancies which require systemic treatment.
17. History of autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medications (other than low dose steroids) within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
To determine recommended phase II dose of human LMY-920 in patients with relapsed or refractory myeloma. | 24 months
  Maximum tolerated dose

SECONDARY OUTCOMES:
To establish toxicity profile for the infusion of LMY-920. | 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. All adverse events during study will be collected, categorized, and graded. Attribution of relatedness to the investigational agent will be assigned.
To determine the objective response rate per International Myeloma Working Group uniform response criteria after treatment with LMY-920 in patients with relapsed or refractory myeloma. | 24 months
  Response rate.
To determine the complete response rate per International Myeloma Working Group uniform response criteria after treatment with LMY-920 in patients with relapsed or refractory myeloma. | 24 months
  Response rate.
To determine the duration of response. | 24 months
  Duration of response
To determine the progression-free survival. | 24 months
  Progression-free survival
To determine the overall survival | 24 months
  Overall survival
To determine incidence of adverse events | 24 months
  Incidence of adverse events
To determine incidence of anti- LMY-920 antibodies | 24 months
  Incidence of anti- LMY-920 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Leland Metheny, MD, Principal Investigator — University Hospitals Seidman Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No